CLINICAL TRIAL: NCT03439033
Title: A Phase 2 Comparison Study of 68Ga-PSMA-HBED-CC Positron Emission Tomography (PET)/CT or PET/MRI Imaging to Magnetic Resonance Imaging (MRI) Alone in Men With Prostate Cancer
Brief Title: Comparison Study of PET/CT or PET/MRI Imaging to Magnetic Resonance Imaging (MRI) Alone in Men With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Drug was FDA approved Summer 2021
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cancer Research & Treatment Fund, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1706018301
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects may be assigned to one of three groups, each with a different intervention in terms of either mode or frequency
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PET/MRI (Experimental): PET/MRI with Gallium-68 labeled PSMA-HBED-CC: Subjects will have one visit during which they will undergo a PET/MRI after being injected with the study drug, Gallium-68 labeled PSMA-HBED-CC.
  Interventions: Drug: PET/MRI with Gallium-68 labeled PSMA-HBED-CC
- Multiple PET/MRI (Experimental): Multiple PET/MRI with Gallium-68 labeled PSMA-HBED-CC: Subjects will be invited to participate in two visits within two years, the second being an optional visit. During each visit, subjects will undergo a PET/MRI after being injected with the study drug, Gallium-68 labeled PSMA-HBED-CC. This arm will be restricted to subjects who plan to undergo focal therapy.
  Interventions: Drug: Multiple PET/MRI with Gallium-68 labeled PSMA-HBED-CC
- PET/CT (Experimental): PET/CT with Gallium-68 labeled PSMA-HBED-CC: Subjects will have one visit during which they will undergo a PET/CT after being injected with the study drug, Gallium-68 labeled PSMA-HBED-CC. PET/CT occurs if a) an MRI can't be performed concurrently; or b) the participant already had an MRI of the abdomen/pelvis or pelvis only.
  Interventions: Drug: PET/CT with Gallium-68 labeled PSMA-HBED-CC

INTERVENTIONS:
Drug: PET/MRI with Gallium-68 labeled PSMA-HBED-CC — Subjects have one visit, during which they will undergo one PET/MRI with the study drug, Gallium-68 labeled PSMA-HBED-CC, a radiopharmaceutical
  Arms: PET/MRI
Drug: Multiple PET/MRI with Gallium-68 labeled PSMA-HBED-CC — Subjects have two visits (the second visit being optional) within two years. During each visit, they will undergo one PET/MRI with the study drug, Gallium-68 labeled PSMA-HBED-CC, a radiopharmaceutical
  Arms: Multiple PET/MRI
Drug: PET/CT with Gallium-68 labeled PSMA-HBED-CC — Subjects have one visit, during which they will undergo one PET/CT with the study drug, Gallium-68 labeled PSMA-HBED-CC, a radiopharmaceutical
  Arms: PET/CT

SUMMARY:
This is a study primarily comparing Magnetic Resonance Imaging (MRI) alone to Positron Emission Tomography (PET)/MRI using an experimental tracer, 68Ga-PSMA-HBED-CC, among men with prostate cancer or prostatic cancer recurrence/metastasis. It is hypothesized that this comparison will demonstrate that PET using the tracer, 68Ga-PSMA-HBED-CC, is more sensitive than MRI alone. Potential subjects who cannot undergo MRI may undergo PET/CT instead.

DETAILED DESCRIPTION:
This is a multi-reader methodological study comparing the diagnostic value of 68Ga-PSMA-HBED-CC PET/CT or 68Ga-PSMA-HBED-CC PET/MRI over MRI alone, using histologic confirmation or serial follow-up for up to 2 years as the gold standard for determination of primary prostate cancer or prostatic cancer recurrence/metastasis. It is hypothesized that this will demonstrate the superiority of 68Ga-PSMA-HBED-CC PET to MRI for sensitivity, and the non-inferiority of 68Ga-PSMA-HBED-CC PET to MRI for specificity.This is a paired, case-control design that is appropriate to statistically evaluate the difference in sensitivity and specificity between the two imaging modalities. Therefore, the estimation of population prevalence is not a study objective, and estimation of clinical utility through calculation of positive and negative predictive values is not appropriate. Imaging studies and follow up subject scans will be organized so that a panel of independent readers will evaluate the MRI and PET studies to assess the level of suspicion for prostate cancer.

ELIGIBILITY:
1. Male aged 21 years or older.
2. Ability to provide signed informed consent and willingness to comply with protocol requirements.
3. Pathologic confirmation of adenocarcinoma of the prostate gland or high clinical suspicion (PSA > 4 ng/mL, or PSA density > 0.15 ng/mL2, or PSA doubling time < 2 years).
4. Meet one of the following 5 criteria

   1. Planned for surgical extirpation, which may or may not include lymph node dissection (high risk primary disease)
   2. Planned for targeted biopsy of primary lesion
   3. Conventional imaging equivocal or suggestive of prostate cancer metastasis/es
   4. Planned focal therapy (with or without radiation therapy) with serial follow-up
   5. Elevated PSA with no conventional imaging suggestive of metastatic or recurrent disease
5. a. If part of PET/MRI cohort, subject will undergo clinically indicated MRI imaging prior to treatment.

   Or b. If part of PET/CT cohort, subject will have had clinically indicated MRI within 3 months prior to treatment.
6. Participants must agree to use an acceptable form of birth control throughout the study period. Participants must use condoms for a period of seven days after each injection, if engaged in sexual activity.

Exclusion Criteria:

1. Clinical and/or technical factors that would compromise statistical analysis of the PET and/or MRI.
2. If part of PET/MRI cohort and patient cohort 3 or 5, subject does not plan to have a prescribed abdomen and pelvis MRI
3. If part of PET/MRI cohort and patient cohort 1, 2 or 4, subject does not plan to have a prescribed pelvis MRI
4. If part of PET/CT cohort and patient cohort 3 or 5, subject does not have previous MR imaging of abdomen and pelvis
5. If part of PET/CT cohort and patient cohort 1, 2 or 4, subject does not have previous MR imaging of pelvis
6. If part of PET/CT cohort, investigator review determines that previous MR images do not meet institutional quality standards
7. If part of PET/MRI cohort, contraindications to MRI
8. Contraindications to PSMA IV administration
9. Other unspecified reasons that, in the opinion of investigators, make the subject unsuitable for enrollment

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Osborne, M.D., Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PSMA PET/MRI Scan vs. MRI Scan: These are males who were referred because of a rising PSA after definitive treatment for prostate cancer. All subjects underwent PSMA PET and MRI from skull base to upper thighs as per convention. Participants received a single IV dose of 4 mCi (148 MBq) +/- 10% of 68Ga-PSMA-HBED-CC (study drug) followed by a PET/MRI scan, 90 min after injection.
Period: Overall Study
Arm/Group | PSMA PET/MRI Scan vs. MRI Scan
Started | 273
Participants With Biochemical Reoccurrence at Baseline | 114
PSMA PET/MRI | 108
PSMA PET/CT | 1
PSMA Multiple PET/MRI | 0
Completed | 109
Not Completed | 164

BASELINE CHARACTERISTICS:
Groups:
- Biochemical Recurrence: These are males who were referred because of a rising PSA after definitive treatment for prostate cancer. All subjects underwent PSMA PET and MRI from skull base to upper thighs as per convention. Participants received a single IV dose of 4 mCi (148 MBq) +/- 10% of 68Ga-PSMA-HBED-CC (study drug) followed by a PET/MRI scan, 90 min after injection.
Arm/Group | Biochemical Recurrence
Number analyzed (Participants) | 114
Age, Continuous [Mean (Full Range); unit: years] | 69 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 114
Stratification Based on PSA Levels [Count of Participants; unit: Participants]
  0 - <0.2 ng/ml | 23
  0.2 <0.5 ng/ml | 33
  0.5 - 2.0 ng/ml | 28
  >2.0 ng/ml | 28
  PSA Levels Unavailable | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Pathologic Lesions Detected by PSMA PET and PET/CT Compared to MP MRI
Description: A scan was considered positive if the clinical interpretation was suspicious based on the clinical judgement of the reader.
Time Frame: At each visit, immediately after administration of the study drug, approximately 2-3 hours; with up to two visits within 2 years or less
Measure: Count of Participants; unit: Participants
Groups:
- PSMA PET/MRI and PET/CT Scan: These are males who were referred because of a rising PSA after definitive treatment for prostate cancer. Patients underwent either PET/MRI or PET/CT. All subjects underwent PSMA PET from skull base to upper thighs as per convention. Participants received a single IV dose of 4 mCi (148 MBq) +/- 10% of 68Ga-PSMA-HBED-CC (study drug) followed by a PET/MRI scan, 90 min after injection.
- MRI Scan: These are males who were referred because of a rising PSA after definitive treatment for prostate cancer. All subjects underwent MRI from skull base to upper thighs as per convention.
Arm/Group | PSMA PET/MRI and PET/CT Scan | MRI Scan
Number analyzed (Participants) | 109 | 109
Participants | 63 | 37

2. Primary Outcome: Number of Pathological Lesions Detected by PSMA PET/MRI and PET/CT Compared to MP MRI in Prostate Cancer Patients With Biochemical Recurrence by Anatomical Region Stratified by PSA Level
Description: Patients were divided into subgroups based on their PSA levels and primary treatment modality. The primary treatment modality subgroups were post radical prostatectomy, post radiation therapy, and post radical prostatectomy and radiation therapy. 109 subjects out of 273 enrolled have data reported. Multiple patients sought care elsewhere and a small number of subjects had 2-year follow-up. This lead to a smaller analysis.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed includes all participants who underwent MRI regardless of whether a pathologic lesion was identified.
Measure: Number; unit: lesions
Arm/Group | PSMA PET/MRI and PET/CT Scan | MRI Scan
Number analyzed (Participants) | 109 | 109
lesions
  Total Number of Lesions | 92 | 47
  PSA Levels 0 to < 0.2 ng/mL | 10 | 0
  PSA Levels 0.2 to < 0.5 ng/mL | 22 | 19
  PSA Levels 0.5 to 2.0 ng/mL | 25 | 10
  PET/MRI: PSA Levels > 2.0 ng/mL | 35 | 18
Statistical Analysis 1: Comparison: PSMA PET/MRI and PET/CT Scan vs MRI Scan; Test type: Superiority; p < 0.0001, McNemar; Risk Difference (RD) = 0.42, 95% CI 2-sided [0.30 to 0.53] — Risk difference reflects PSMA PET/MRI Scan detection proportion minus MRI scan detection proportion

3. Secondary Outcome: Number of Pathological Lesions Detected by PSMA PET/MRI and PET/CT Compared to MP MRI in Prostate Cancer Patients With Biochemical Recurrence by Anatomical Region
Description: True positive rates for detecting lesions between PSMA PET/MRI and MP MRI in various anatomical locations were compared, including prostate/prostatic bed, N1 lymph nodes, N2 lymph nodes, and osseous lesions. Other anatomical sites are other than bone, node, and prostate.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: lesions
Arm/Group | PSMA PET/MRI and PET/CT Scan | MRI Scan
Number analyzed (Participants) | 109 | 109
lesions
  Total Number of Lesions | 92 | 47
  N1 lymph nodes | 34 | 11
  N2 lymph nodes | 20 | 7
  Osseous | 24 | 14
  Prostate | 3 | 7
  Prostatic Bed | 8 | 7
  Other Anatomical Sites | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected after each visit (approximately 1-3 hours), immediately post-scan and up to 2 years post-scan.
Description: This study follows standard operating procedures for reporting adverse events and utilize the AE grading from Common Terminology Criteria for Adverse Events v4.0.
Groups:
- PSMA PET/MRI Scan; MRI Scan: These are males who were referred because of a rising PSA after definitive treatment for prostate cancer. All subjects underwent PSMA PET and MRI from skull base to upper thighs as per convention. Participants received a single IV dose of 4 mCi (148 MBq) +/- 10% of 68Ga-PSMA-HBED-CC (study drug) followed by a PET/MRI scan, 90 min after injection.
- PSMA PET/CT: PET/CT with Gallium-68 labeled PSMA-HBED-CC: Subjects will have one visit during which they will undergo a PET/CT after being injected with the study drug, Gallium-68 labeled PSMA-HBED-CC. PET/CT occurs if a) an MRI can't be performed concurrently; or b) the participant already had an MRI of the abdomen/pelvis or pelvis only.
- PSMA Multiple PET/MRI: Multiple PET/MRI with Gallium-68 labeled PSMA-HBED-CC: Subjects will be invited to participate in two visits within two years, the second being an optional visit. During each visit, subjects will undergo a PET/MRI after being injected with the study drug, Gallium-68 labeled PSMA-HBED-CC. This arm will be restricted to subjects who plan to undergo focal therapy.
Arm/Group | PSMA PET/MRI Scan | MRI Scan | PSMA PET/CT | PSMA Multiple PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/273 | 0/273 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/273 | 0/273 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/273 | 0/273 | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
One limitation is the small number of cases available for specificity analysis resulting in a negligible sample size of patients who had a true negative reference. Another limitation is multiple patients sought care at other institutions. As a result, information was not complete for several patients. Only a small number of the subjects had 2-year follow-up or underwent confirmatory biopsy, which introduces the possibility of selection bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT03439033/Prot_SAP_000.pdf